CLINICAL TRIAL: NCT05955066
Title: Effect of JAK Inhibitor on Bone Erosion Repair in Rheumatoid Arthritis Assessed by HR-pQCT: a Randomized Placebo-controlled Study
Brief Title: Effect of JAK Inhibitor on Erosion Healing in RA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ho SO, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JAKi
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib (Experimental): Patients randomized into JAKi group will receive one capsule of baricitinib (4mg) daily for 24 weeks.
  Interventions: Drug: Baricitinib 4 MG
- Placebo (Placebo Comparator): Patients randomized into placebo group will receive one capsule of placebo daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib 4 MG — 1 capsule (4mg) daily for 24 weeks
  Other Names: Olumiant
  Arms: Baricitinib
Drug: Placebo — 1 capsule daily
  Arms: Placebo

SUMMARY:
Objective To investigate the effect of Janus kinase (JAK) inhibition by baricitinib on erosion healing in rheumatoid arthritis (RA) patients with active disease using high-resolution peripheral quantitative computer tomography(HR-pQCT).

Hypothesis JAK inhibitor can lead to healing of existing erosion in RA patients with active disease.

Design and subjects This is a 24-week, randomized, placebo-controlled, double-blind study. We plan to enroll 60 adult patients with active RA (Disease activity score 28-C-reactive protein [DAS28-CRP]>3.2) and 1 bone erosion on HR-pQCT. They will be randomized 1:1 to receive JAK inhibitor (baricitinib 4mg once daily) or placebo for 24 weeks. Medications will be adjusted according to a standard protocol aiming to achieve low disease activity. Patients requiring biologic or other targeted synthetic disease-modifying-anti-rheumatic-drugs will be excluded.

Study instruments HR-pQCT of the 2-4 metacarpophalangeal(MCP) will be done at baseline and 24 weeks. Inflammatory cytokine profile and bone cartilage interface biomarkers will also be checked at baseline and 24 weeks. Clinical response will be monitored using DAS28-CRP.

Main outcome measures and analysis The primary outcome is the proportion of patients with erosion volume regression on HR-pQCT comparing the two groups by chisquare test.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a common chronic inflammatory arthritis affecting 0.35% of the population in Hong Kong. Uncontrolled arthritis can lead to joint destruction, functional disability and decreased quality of life. We also found that the disease carried substantial socioeconomic costs.

Bone erosions are specific to RA reflecting disease severity, and can be used to monitor disease progression. In early RA, functional capacity is most associated with disease activity, but in established disease, with joint damage. A recent study also showed joint tenderness, a crucial determinant of disease activity, was associated with structural damage rather than sonographic synovitis in non-swollen joints in established RA. In fact, prevention of erosion on radiographs is used to define the efficacy of disease modifying anti-rheumatic drugs (DMARDs) in RA. After all, the ultimate aims of management in RA are to reduce symptoms, preserve function and maintain quality of life.

The 60 patients with erosion will be randomized in a 1:1 ratio to JAK1 inhibitor (n=30) or placebo (n=30) group. Randomization will be performed using a computer-generated randomization list provided by the research pharmacist, using a permuted blocks design with block sizes of 4. Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes. Treatment will be masked to patients and investigators.

All the participants will be instructed to take one study capsule (4 mg baricitinib or placebo) daily for 24 weeks. They will be treated to the target of DAS28 remission or low disease activity (LDA) at PWH throughout the study period according to a standard protocol modified to our study based on the EULAR recommendation and the Hong Kong guideline on the use of DMARDs. Disease activity and adverse events will be monitored at 4 weeks, 12 weeks and 24 weeks. Patients will be advised to reach out to the rheumatologists earlier if the condition changes unexpectedly. Changes in treatment, e.g. the switching to a new csDMARD including leflunomide, hydroxychloroquine, or sulfasalazine or the dosage of csDMARDs and changes in the dosage or the addition of glucocorticoids or nonsteroidal anti-inflammatory drugs are allowed throughout the study. The use of b/tsDMARDs, bisphosphonates, denosumab, teriparatide or systemic glucocorticoid > prednisolone 10 mg/day equivalent will be prohibited throughout the study. Participants who required rescue b/tsDMARDs will be withdrawn from the study and excluded from the final analysis.

The following clinical variables will be assessed at each visit: erythrocyte sedimentation rate (ESR), CRP, number of swollen joints (0-28), number of tender joints (0-28), visual analogue scale (VAS) for pain (0-100 mm=most pain), VAS for patient's global assessment (0-100 mm=worst score), VAS for physician's global assessment (0-100 mm=worst score), and DAS28 score. The number of damaged joints will be assessed at baseline and the end of the study. Rheumatoid factor status and anti-cyclic citrullinated peptide antibodies status will be determined at baseline. Functional disability is assessed by the disability index of HAQ (0-3=most functional disability). ACR20/50/70 responses are defined as at least 20%, 50%, and 70% improvement in swollen joint and tender joint counts, and three of five other variables (i.e., ESR or CRP, HAQ score, pain score, and physicians' and patients' global assessments).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 year-old,
2. fulfilment of the 2010 ACR/EULAR classification criteria of RA,
3. on MTX for at least 12 weeks, and
4. disease activity score 28-C-reactive protein (DAS28-CRP) > 3.2.

Exclusion Criteria:

1. ≥65 years old,
2. functional status class IV (limited in ability to perform usual self-care, vocational, and avocational activities);
3. pregnancy or premenopausal women planning pregnancy;
4. ever use of any b/tsDMARDs or csDMARDs other than methotrexate and hydroxychloroquine for RA;
5. ever use of bisphosphonates, denosumab or teriparatide;
6. history of cardiovascular disease/thrombo-embolism/malignancy;
7. contraindications to baricitinib; and
8. severe joint damage in MCP2-4 which preludes HR-pqCT measurement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with reduction of erosion volume on HR-pQCT over 2-4 metacarpophalangeal (MCP 2-4) at 24 weeks comparing JAK inhibitor group and placebo group. | 24 weeks
  Bone erosion will be assessed at MCP 2-4 of the most affected hand or dominant hand when both hands are equally affected.
  The primary outcome measurement, the comparison of proportion of patients with erosion volume reduction in the 2 groups, will be analyzed by the Chi-square test. Clinical variables which are significantly different between the 2 groups in the univariate analyses and are biologically plausible (eg. age, sex, disease duration, disease activity or treatment) will be adjusted in the multivariate logistic regression model to confirm the JAK inhibitor treatment effect.

SECONDARY OUTCOMES:
The proportion of patients with definitive erosion healing on HR-pQCT at 24 weeks comparing the 2 groups, with definite erosion defined as 1) a decrease in erosion volume exceeding the smallest | 24 weeks
  Bone erosion will be assessed at MCP 2-4 of the most affected hand or dominant hand when both hands are equally affected.
  The secondary outcome on definitive erosion healing will be compared likewise. To address the secondary outcomes on changes of erosion parameters, disease activity and biomarkers, the comparison will be done by T-test or Mann-Whitney U test. The within group changes of these measurements before and after treatment will be examined using paired t-test or Wilcoxon signed-rank test. Independent factors predicting treatment response in the JAK inhibitor group will be analyzed by multivariate logistic regression. A 2-tailed probability value of p<0.05 is considered statistically significant.
Changes in dimensions of erosion (depth, width and volume), marginal osteosclerosis and joint space width (minimal, maximal, asymmetry and distribution) on HR-pQCT at 24 weeks comparing the 2 groups. | 24 weeks
  Bone erosion will be assessed at MCP 2-4 of the most affected hand or dominant hand when both hands are equally affected.
  The secondary outcome on definitive erosion healing will be compared likewise. To address the secondary outcomes on changes of erosion parameters, disease activity and biomarkers, the comparison will be done by T-test or Mann-Whitney U test. The within group changes of these measurements before and after treatment will be examined using paired t-test or Wilcoxon signed-rank test. Independent factors predicting treatment response in the JAK inhibitor group will be analyzed by multivariate logistic regression. A 2-tailed probability value of p<0.05 is considered statistically significant.
Changes in RA disease activity at 24 weeks comparing the 2 groups. | 24 weeks
  Disease activity and adverse events will be monitored at 4 weeks, 12 weeks and 24 weeks. The following clinical variables will be assessed at each visit: erythrocyte sedimentation rate (ESR), CRP, number of swollen joints (0-28), number of tender joints (0-28), visual analogue scale (VAS) for pain (0-100 mm=most pain), VAS for patient's global assessment (0-100 mm=worst score), VAS for physician's global assessment (0-100 mm=worst score), and DAS28 score. The number of damaged joints will be assessed at baseline and the end of the study. Rheumatoid factor status and anti-cyclic citrullinated peptide antibodies status will be determined at baseline. Functional disability is assessed by the disability index of HAQ (0-3=most functional disability).
Changes in the inflammatory cytokines/chemokines and bone-cartilage biomarkers comparing the 2 groups. | 24 weeks
  Bone erosion will be assessed at MCP 2-4 of the most affected hand or dominant hand when both hands are equally affected.
  The secondary outcome on definitive erosion healing will be compared likewise. To address the secondary outcomes on changes of erosion parameters, disease activity and biomarkers, the comparison will be done by T-test or Mann-Whitney U test. The within group changes of these measurements before and after treatment will be examined using paired t-test or Wilcoxon signed-rank test. Independent factors predicting treatment response in the JAK inhibitor group will be analyzed by multivariate logistic regression. A 2-tailed probability value of p<0.05 is considered statistically significant.
Predictors of response to JAK inhibitor treatment in terms of erosion healing. | 24 week
  The secondary outcome on definitive erosion healing will be compared likewise. To address the secondary outcomes on changes of erosion parameters, disease activity and biomarkers, the comparison will be done by T-test or Mann-Whitney U test. The within group changes of these measurements before and after treatment will be examined using paired t-test or Wilcoxon signed-rank test. Independent factors predicting treatment response in the JAK inhibitor group will be analyzed by multivariate logistic regression. A 2-tailed probability value of p<0.05 is considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized clinical data can be shared upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the final manuscript
Access Criteria: For research purpose